CLINICAL TRIAL: NCT04117425
Title: Study of Maternal Pharmacokinetic and Placental Transfer of Levetiracetam
Brief Title: Pharmacokinetic and Placental Transfer of Levetiracetam
Acronym: EPICEINTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRC17036
Record Dates: First submitted 2019-06-04; First posted 2019-10-07 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy in Pregnancy
Keywords: Epilepsy; pharmacokinetic; levetiracetam; placental transfer.
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Protocol to determine the optimal dose of levetiracetam during pregnancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Other): 40 Pregnant women and 10 Pregnant women that have a medical interruption of pregnancy who were already treated by levetiracetam.
  Blood collection at each trimester of pregnancy, delivery and post partum visit or at medical interruption.
  Collection of saliva at each trimester of pregnancy and post partum visit. Collection of cord blood and amniotic fluid at delivery or at medical interruption
  Interventions: Biological: biological collection

INTERVENTIONS:
Biological: biological collection — Blood collection at each trimester of pregnancy, delivery and post partum visit or at medical interruption.
  Collection of saliva at each trimester of pregnancy and post partum visit. Collection of cord blood and amniotic fluid at delivery or at medical interruption.

SUMMARY:
Hypotheses: The treatment of epilepsy during pregnancy is difficult because of the risk of anti-epileptic drugs on the one hand and the risk of destabilization of epilepsy in the mother on the other hand. There is limited data on the pharmacokinetics (concentration study) and pharmacodynamics (efficacy and toxicity effects study) of levetiracetam in pregnant women. The few studies focus on few women and show very strong interindividual variability and a tendency to decrease total concentrations.

Main objective: To develop a population pharmacokinetic model of levetiracetam during pregnancy. After the study, this model could be used to propose dose adjustments to maintain stable concentrations in pregnant women throughout pregnancy.

Secondary objectives:

* Describe placental transfer during childbirth and during a medical termination of pregnancy
* Link the concentration and its variation in the individual to the effects of treatment

DETAILED DESCRIPTION:
Methodology: Are included by the neurology service, pregnant women which are already under levetiracetam and / or obstetric gynecology services for her treatment of epilepsy, pregnant women at first consultation. Women are already taking levetiracetam and the drug is not provided by the study40 mother-child couples, as well as 10 women who undergo a medical termination of pregnancy will have to be included in the study, in 7 maternities in Paris.

Women are already taking the drugs, according to the practices of the different services, and the study will not change their prescriptions of these drugs. The women will have a blood sample at 3 visits during pregnancy (11-14 weeks, 24-28 weeks and 35-39 weeks) and at the post-partum consultation. At delivery, a collection of the mother, cord blood and amniotic fluid will be performed. A salivary specimen will be routinely collected at the same time as the mother's plasma sample.

The pharmaco-statistical analysis will be conducted using non-linear mixed-effect modeling programs (Monolix and Nonmem) to calculate the main pharmacokinetic parameters of the mother and fetus and to estimate their variability. This type of modeling makes it possible to take into account individual covariates (weight, gestational age ...) to explain the pharmacokinetic variability between mother - child pairs. The final model will be validated by a simulation technique. The final model will be used to rationalize the changes in antiepileptic doses during pregnancy and to explain the differences in passage, based on individual covariates, then to perform simulations to find out how to modify the administration for treatment to be effective as often as possible.

The secondary endpoints are

* Exposure ratio (area under the concentration-time curve) between the mother and the fetus to describe the transplacental passage of levetiracetam levetiracetam.
* To correlate the evolution of the concentrations in the woman (value in the woman whose treatment is balanced before the pregnancy minus the value when she is pregnant) to

  * the effectiveness (number of crises that the patient did).
  * tolerance: presence or absence of clinical and biological abnormalities occurring in pregnant women and children

ELIGIBILITY:
Inclusion Criteria:

* pregnant Women of childbearing age who are pregnant
* Age ≥18 years
* Women with epilepsy treated with levetiracetam in monotherapy or combination
* affiliated to a social security scheme (or entitled)

Exclusion Criteria:

* Women treated with antiepileptics for pathology other than epilepsy
* Women treated with a combination of more than 3 antiepileptics
* Severe anemia
* Renal failure (moderate to severe)
* Hepatic impairment (moderate to severe)
* Alcohol and/or recreational drug use
* Trend towards non-compliance with treatment
* Inability to maintain a Crisis Observation Workbook
* Suicidal Ideas
* Uncontrolled thyroid disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Levetiracetam pharmacokinetics in pregnancy | At delivery
  Levetiracetam concentrations as a function of time

SECONDARY OUTCOMES:
Levetiracetam pharmacokinetics in pregnancy | At inclusion
  Levetiracetam concentrations as a function of time
Levetiracetam pharmacokinetics in pregnancy | Until 17 weeks
  Levetiracetam concentrations as a function of time
Levetiracetam pharmacokinetics in pregnancy | Until 28 weeks
  Levetiracetam concentrations as a function of time
Levetiracetam pharmacokinetics in pregnancy | Until 6 week after delivery
  Levetiracetam concentrations as a function of time
Exposure ratio | At delivery
  area below the concentration curve as a function of time) between the mother and the fetus to describe the transplacental passage of levetiracetam.
Link between levetiracetam concentrations and effects | At inclusion
  correlate the evolution of the concentrations in the woman (value in the woman whose treatment is balanced before the pregnancy minus the value when she is pregnant) to
  * the effectiveness (number of crises that the patient did).
  * tolerance: presence or absence of clinical and biological abnormalities occurring in pregnant women and children.
Link between levetiracetam concentrations and effects | Until 17 weeks
  Correlate the evolution of the concentrations in the woman (value in the woman whose treatment is balanced before the pregnancy minus the value when she is pregnant) to
  * the effectiveness (number of crises that the patient did).
  * tolerance: presence or absence of clinical and biological abnormalities occurring in pregnant women and children
Link between levetiracetam concentrations and effects | Until 28 weeks
  Correlate the evolution of the concentrations in the woman (value in the woman whose treatment is balanced before the pregnancy minus the value when she is pregnant) to
  * the effectiveness (number of crises that the patient did).
  * tolerance: presence or absence of clinical and biological abnormalities occurring in pregnant women and children
Link between levetiracetam concentrations and effects | Until 6 week after delivery
  Correlate the evolution of the concentrations in the woman (value in the woman whose treatment is balanced before the pregnancy minus the value when she is pregnant) to
  * the effectiveness (number of crises that the patient did).
  * tolerance: presence or absence of clinical and biological abnormalities occurring in pregnant women and children.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Tréluyer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- hospital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pennell PB. Antiepileptic drug pharmacokinetics during pregnancy and lactation. Neurology. 2003 Sep 1;61(6 Suppl 2):S35-42. doi: 10.1212/wnl.61.6_suppl_2.s35. PMID 14504308
- [Background] Tomson T, Palm R, Kallen K, Ben-Menachem E, Soderfeldt B, Danielsson B, Johansson R, Luef G, Ohman I. Pharmacokinetics of levetiracetam during pregnancy, delivery, in the neonatal period, and lactation. Epilepsia. 2007 Jun;48(6):1111-6. doi: 10.1111/j.1528-1167.2007.01032.x. Epub 2007 Mar 22. PMID 17381438
- [Background] Westin AA, Reimers A, Helde G, Nakken KO, Brodtkorb E. Serum concentration/dose ratio of levetiracetam before, during and after pregnancy. Seizure. 2008 Mar;17(2):192-8. doi: 10.1016/j.seizure.2007.11.027. Epub 2008 Jan 3. PMID 18180176